CLINICAL TRIAL: NCT03595891
Title: Apixaban Length-Of-Stay Pulmonary Embolism Study - Hospital Admissions (ALPHA-PE)
Brief Title: The Study of How Long Participants Stay in the Hospital After Receiving Apixaban for a Blood Clot in the Lung
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-640
Record Dates: First submitted 2018-05-08; First posted 2018-07-23 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Embolism (PE); Pulmonary Thromboembolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult with acute PE before the introduction of apixaban
  Interventions: Other: Non-Interventional
- Adult with acute PE after the introduction of apixaban
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
A study based on a chart review of participants that presented with a sudden blood clot in the lung

ELIGIBILITY:
Inclusion Criteria:

* Adults participants at date of admission
* Primary presentation consistent with PE followed by objectively-confirmed acute PE
* Received anti-coagulation upon diagnosis of PE during study period and in receipt of anti-coagulation at discharge

Exclusion Criteria:

* PE diagnosed during a hospital admission for a reason other than PE during the study period
* Patients receiving anticoagulation at the time of presentation
* Patients presenting outside the defined study period

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years of age) at index date presenting with acute Pulmonary Embolism (PE), which was then objectively confirmed, and received anticoagulation upon diagnosis of PE and in receipt of anticoagulation at discharge.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Compare the average length of stay in secondary care | 60 days

SECONDARY OUTCOMES:
Total length of stay, including repeat admissions | During the first 30 days after presentation of PE
Distribution of clinical characteristics of patients admitted with a PE | Baseline
  Clinical characteristics will be summarized using descriptive statistics
Distribution of demographic data of patients admitted with a PE | Baseline
  Demographic data will be summarized using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Cardiff, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm